CLINICAL TRIAL: NCT05431348
Title: Effect of StRess and ExeRcize on the Outcome After Chemo-Radiation
Acronym: ERROR
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ERROR
Record Dates: First submitted 2022-02-22; First posted 2022-06-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma (GBM)
Keywords: stress; glioblastoma; survival; quality of life
MeSH Terms: conditions — Glioblastoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with glioblastoma treated with STUPP schema
  Interventions: Device: Smartwatch; Diagnostic Test: Serum Cortisol; Other: Questionnaires

INTERVENTIONS:
Device: Smartwatch — Patients will wear the smartwatch during treatment which measures, activity, steps, sleep and heartrate
Diagnostic Test: Serum Cortisol — Level of cortisol in serum will be determined
Other: Questionnaires — Patients are asked to fill in patient reported outcomes (PROMS) and specific questions on stress, exercise and fatigue (QSC-R23, IPAQ-SF, MVI-20)

SUMMARY:
Glioblastoma (GBM) is a highly malignant, incurable primary brain tumor. Due to the nature of this disease and the extent of the treatment (surgery followed by chemoradiation according to the Stupp trial) patients undergo considerable psychological distress. It is known that stress hormones are involved in a wide range of processes involved in cell survival, cell cycle and immune function, and can cause therapy resistance. In this study the effect of stress on outcome after chemoradiation in patients with GBM will be investigated.

DETAILED DESCRIPTION:
Psychological stress will be measured using multiple approaches; Physiological measures, stress biomarker and questionnaires. Using this approach, a broad insight in the relationship between stress and outcome after chemoradiation will be obtained and the potential influence of physical activity and sleep evaluated. In addition, the results of this study will help to identify patients which experience high stress levels during chemoradiation to pilot (in the future) interventions to reduce stress before and during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Stupp or Elderly protocol: GBM WHO IV, astrocytoma WHO IV IDHmt, astrocytoma WHO II IDHwt (GBM-like).
* willing to wear the smart watch during the treatment protocol

Exclusion Criteria:

* younger than 18 years
* not in possession of a smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a glioblastoma (GBM) eligible for treatment with STUPP or Elderly treatment protocol (concurrent radio-chemotherapy + temozolomide)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Is stress a prognostic factor for the overall survival of patients with glioblastoma (GBM)? | 1 year
  Stress variables are heartrate (min, max, average), sleep (duration, interruptions), serum cortisol and Questionnaire on Stress in Cancer Patients revised version (QSC-23) are related to overall survival at 1 year (survival = yes/no)
Is stress a prognostic factor for the progression free- survival at 1 year of patients with glioblastoma (GBM)? | 1 year
  Stress variables are heartrate (min, max, average), sleep (duration, interruptions), serum cortisol and Questionnaire on Stress in Cancer Patients revised version (QSC-23) are related to progression free survival at 1 year (progression free survival at 1 year; yes/no)

SECONDARY OUTCOMES:
Is stress a prognostic factor for the quality of life of patients with GBM | 1 year
  Stress variables like heartrate, sleep, serum cortisol and the Questionnaire on Stress in Cancer Patients revised version (QSC-23) are related to quality of life (EuroQol 5D)
  EuroQol 5D: The 5 questions on the health condition will be scored on a 3-point scale (1-3) By placing these numbers after each other a 5-digit index will occur which provides the health profile. This 5-digit number can be re-calculated to a total score.
Is stress a prognostic factor for dose limiting toxicities (CTC) of the treatment? | 1 year
  Stress variables like heartrate (min, max, average), sleep (duration, interruptions), serum cortisol and Questionnaire on Stress in Cancer Patients revised version (QSC-23) are related to EORTC Common Toxicity Criteria (CTC) score.
  CTC: ranging from grade 1: mild to 5: death
Is stress a prognostic factor for early termination of the treatment? | 1 year
  Stress variables like heartrate (min, max, average), sleep (duration, interruptions), serum cortisol and Questionnaire on Stress in Cancer Patients revised version (QSC-23) are related to early treatment cessation.
  early treatment cessation (yes/no)
Is there a relationship between stress and treatment response measures on MRI imaging | 6 months
  Stress variables like heartrate (min, max, average), sleep (duration, interruptions), serum cortisol and Questionnaire on Stress in Cancer Patients revised version (QSC-23) are related to potential changes in clinical MRI (clinical significant edema and/or clinical significant radionecrosis)
  Potential changes in clinical MRI (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zegers, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastricht Radiation Oncology (Maastro), Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Zabora J, BrintzenhofeSzoc K, Curbow B, Hooker C, Piantadosi S. The prevalence of psychological distress by cancer site. Psychooncology. 2001 Jan-Feb;10(1):19-28. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-6. PMID 11180574
- [Background] Sehlen S, Hollenhorst H, Schymura B, Herschbach P, Aydemir U, Firsching M, Duhmke E. Psychosocial stress in cancer patients during and after radiotherapy. Strahlenther Onkol. 2003 Mar;179(3):175-80. doi: 10.1007/s00066-003-1018-z. PMID 12627260
- [Background] Kelly C, Majewska P, Ioannidis S, Raza MH, Williams M. Estimating progression-free survival in patients with glioblastoma using routinely collected data. J Neurooncol. 2017 Dec;135(3):621-627. doi: 10.1007/s11060-017-2619-1. Epub 2017 Sep 27. PMID 28956223
- [Background] Mattern J, Buchler MW, Herr I. Cell cycle arrest by glucocorticoids may protect normal tissue and solid tumors from cancer therapy. Cancer Biol Ther. 2007 Sep;6(9):1345-54. doi: 10.4161/cbt.6.9.4765. Epub 2007 Jul 19. PMID 18087223